CLINICAL TRIAL: NCT05419531
Title: Measuring the Incidence of Colorectal Cancer in Young Endurance Athletes
Brief Title: The Purpose of This Study is to Determine the Frequency of Colorectal Cancer in Male and Female Endurance Athletes Between the Ages of 35 and 50
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: U21-10-4567
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prospective observational study - screening and follow up colonoscopy — Involves two visits and a colonoscopy. The first visit will be prior to the colonoscopy. 4-35 days after the colonoscopy, there will be a one time appointment to go over the results of the colonoscopy.

SUMMARY:
The purpose of this study is to determine the frequency of colorectal cancer in male and female endurance athletes between the ages of 35 and 50.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females 35-50 years of age
* Male and female self-reported endurance athletes, defined by at least one of the following:

  * Run at least two races of 50 miles or more
  * Run 5 races of 26.2 miles or more
* Ability to complete testing in the protocol and make study visits
* Able and willing to consent to protocol

Exclusion Criteria:

* Known or suspected history of inflammatory bowel disease, familial adenomatous polyposis (FAP), or Lynch Syndrome
* Concomitant illness that would prevent adequate patient assessment or in the investigators' opinion pose an added risk for study participants.
* Anticipated poor compliance
* Prisoners or subjects who are involuntarily incarcerated
* Persons with decisional incapacity/cognitive impairment
* Any history or evidence of severe illness or any other condition that would make the patient, in the opinion of the investigator unsuitable for the study
* Subject is involved with a worker's compensation, personal injury, or other legal matters related to their health
* Subject is enrolled in a separate interventional clinical trial

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Potential participants will be recruited through distribution of a flyer at endurance events, chat rooms, and race invitations.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
The rate of young endurance runners' that have adenomatous polyps. | 36 months
  1. Estimate the rate of young endurance runners that have adenomatous polyps.
  2. Estimate the rate of young endurance runners that have advanced adenoma and colorectal cancer on screening colonoscopies.

SECONDARY OUTCOMES:
Comparison of the rate of young endurance athletes that have adenomatous polyps with that of the historical controls (those in the average risk group). | 36 months
  Fisher's Exact test will be used to compare the rates of adenomatous polyps and colorectal cancer between the young endurance athletes and that of the historical controls.
  2.3 Secondary Objectives
  1. Compare the rate of young endurance runners that have adenomatous polyps with that of the historical controls (those in the average risk group)
  2. Compare the rate of young endurance runners that have advanced adenoma and colorectal cancer on screening colonoscopies with that of the historical controls (those in the average risk group).
Comparison of the rate of young endurance athletes that have colorectal cancer on screening colonoscopies with that of the historical controls (those in the average risk group). | 36 months
  Fisher's Exact test will be used to compare the rates of adenomatous polyps and colorectal cancer between the young endurance athletes and that of the historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cannon, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Fedewa SA, Anderson WF, Miller KD, Ma J, Rosenberg PS, Jemal A. Colorectal Cancer Incidence Patterns in the United States, 1974-2013. J Natl Cancer Inst. 2017 Aug 1;109(8):djw322. doi: 10.1093/jnci/djw322. PMID 28376186
- [Background] Meyer JE, Narang T, Schnoll-Sussman FH, Pochapin MB, Christos PJ, Sherr DL. Increasing incidence of rectal cancer in patients aged younger than 40 years: an analysis of the surveillance, epidemiology, and end results database. Cancer. 2010 Sep 15;116(18):4354-9. doi: 10.1002/cncr.25432. PMID 20734460
- [Background] Cong YJ, Gan Y, Sun HL, Deng J, Cao SY, Xu X, Lu ZX. Association of sedentary behaviour with colon and rectal cancer: a meta-analysis of observational studies. Br J Cancer. 2014 Feb 4;110(3):817-26. doi: 10.1038/bjc.2013.709. Epub 2013 Nov 21. PMID 24263062
- [Background] Heer M, Repond F, Hany A, Sulser H, Kehl O, Jager K. Acute ischaemic colitis in a female long distance runner. Gut. 1987 Jul;28(7):896-9. doi: 10.1136/gut.28.7.896. PMID 3498668
- [Background] Sanchez LD, Tracy JA, Berkoff D, Pedrosa I. Ischemic colitis in marathon runners: a case-based review. J Emerg Med. 2006 Apr;30(3):321-6. doi: 10.1016/j.jemermed.2005.05.021. PMID 16677987
- [Background] Casey E, Mistry DJ, MacKnight JM. Training room management of medical conditions: sports gastroenterology. Clin Sports Med. 2005 Jul;24(3):525-40, viii. doi: 10.1016/j.csm.2005.05.002. PMID 16004918
- [Background] de Oliveira EP, Burini RC. The impact of physical exercise on the gastrointestinal tract. Curr Opin Clin Nutr Metab Care. 2009 Sep;12(5):533-8. doi: 10.1097/MCO.0b013e32832e6776. PMID 19535976
- [Background] Clausen JP. Effect of physical training on cardiovascular adjustments to exercise in man. Physiol Rev. 1977 Oct;57(4):779-815. doi: 10.1152/physrev.1977.57.4.779. No abstract available. PMID 333481
- [Background] Kehl O, Jager K, Munch R, Buhler H, Segantini P, Bollinger A, Ammann R. [Mesenterial anemia as a cause of jogging anemia?]. Schweiz Med Wochenschr. 1986 Jul 19;116(29):974-6. German. PMID 3764381
- [Background] Porter AM. Do some marathon runners bleed into the gut? Br Med J (Clin Res Ed). 1983 Nov 12;287(6403):1427. doi: 10.1136/bmj.287.6403.1427. No abstract available. PMID 6416441
- [Background] Baska RS, Moses FM, Graeber G, Kearney G. Gastrointestinal bleeding during an ultramarathon. Dig Dis Sci. 1990 Feb;35(2):276-9. doi: 10.1007/BF01536777. PMID 2302987
- [Background] Blokzijl F, de Ligt J, Jager M, Sasselli V, Roerink S, Sasaki N, Huch M, Boymans S, Kuijk E, Prins P, Nijman IJ, Martincorena I, Mokry M, Wiegerinck CL, Middendorp S, Sato T, Schwank G, Nieuwenhuis EE, Verstegen MM, van der Laan LJ, de Jonge J, IJzermans JN, Vries RG, van de Wetering M, Stratton MR, Clevers H, Cuppen E, van Boxtel R. Tissue-specific mutation accumulation in human adult stem cells during life. Nature. 2016 Oct 13;538(7624):260-264. doi: 10.1038/nature19768. Epub 2016 Oct 3. PMID 27698416
- [Background] Tomasetti C, Li L, Vogelstein B. Stem cell divisions, somatic mutations, cancer etiology, and cancer prevention. Science. 2017 Mar 24;355(6331):1330-1334. doi: 10.1126/science.aaf9011. PMID 28336671
- [Background] Scott JP, Sale C, Greeves JP, Casey A, Dutton J, Fraser WD. Effect of exercise intensity on the cytokine response to an acute bout of running. Med Sci Sports Exerc. 2011 Dec;43(12):2297-306. doi: 10.1249/MSS.0b013e31822113a9. PMID 21552156
- [Background] Nieman DC, Konrad M, Henson DA, Kennerly K, Shanely RA, Wallner-Liebmann SJ. Variance in the acute inflammatory response to prolonged cycling is linked to exercise intensity. J Interferon Cytokine Res. 2012 Jan;32(1):12-7. doi: 10.1089/jir.2011.0038. Epub 2011 Sep 14. PMID 21916608
- [Background] Xu G, Lin W, McAinch AJ, Yan X, Weng X. Identification of Urinary Biomarkers for Exercise-Induced Immunosuppression by iTRAQ Proteomics. Biomed Res Int. 2020 Jan 23;2020:3030793. doi: 10.1155/2020/3030793. eCollection 2020. PMID 32047808
- [Background] Thomas RJ, Kenfield SA, Jimenez A. Exercise-induced biochemical changes and their potential influence on cancer: a scientific review. Br J Sports Med. 2017 Apr;51(8):640-644. doi: 10.1136/bjsports-2016-096343. Epub 2016 Dec 19. PMID 27993842
- [Background] Steiner P. When suspected 'runner's colitis' in a marathon runner turns out to be cancer-and in the end leads to a new personal best marathon time. Br J Sports Med. 2020 Mar;54(5):311-312. doi: 10.1136/bjsports-2019-100675. Epub 2019 Aug 2. No abstract available. PMID 31375499
- [Background] Hemmasi G, Sohrabi M, Zamani F, Ajdarkosh H, Rakhshani N, Khoonsari M, Ameli M, Hatami K. Prevalence of colorectal adenoma in an average-risk population aged 40-50 versus 50-60 years. Eur J Cancer Prev. 2015 Sep;24(5):386-90. doi: 10.1097/CEJ.0000000000000097. PMID 25380192